CLINICAL TRIAL: NCT07012798
Title: A Prospective, Single-arm, Single-center Phase II Clinical Study of Hepatic Artery Infusion Chemotherapy (FOLFOX) Combined With Durvalumab (MEDI4736), Bevacizumab, and Stereotactic Body Radiotherapy in Sequential Treatment of Potentially Resectable Locally Advanced Hepatocellular Carcinoma
Brief Title: FOLFOX Combined With Durvalumab (MEDI4736), Bevacizumab, and Stereotactic Body Radiotherapy in Sequential Treatment of Potentially Resectable Locally Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB-HERO
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Durvalumab; HAIC; SBRT; Conversion Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TREATMENT (Experimental): therapy of durvalumab in combination with bevacizumab, combined with HAIC followed by SBRT
  Interventions: Drug: Durvalumab; Drug: Bevacizumab; Drug: HAIC of FOLFOX

INTERVENTIONS:
Drug: Durvalumab — 1120mg, iv, q3w
Drug: Bevacizumab — 15mg/kg, iv, q3w
Drug: HAIC of FOLFOX — HAIC (FOLFOX): oxaliplatin 100mg/m2, 4h, day 1 + leucovorin 300mg/m2, 2h, day
  1 + fluorouracil 500mg/m2, 20min, day 1 + fluorouracil 1500mg/m2, 20h, q3w

SUMMARY:
Study Design:

This is a pilot study with a single arm in a single centre assessing safety and efficacy of durvalumab in combination with bevacizumab and HAIC followed by SBRT. This study will be conducted in selected patients with intermediate or advanced stage HCC not amenable to curative therapy. Approximately 30 patients will be enrolled and receive treatments.

Primary Objectives:

To evaluate the possibility of HAIC plus durvalumab and bevacizumab followed by SBRT as conversion therapy for HCC.

Secondary Objective(s):

To evaluate the efficacy of HAIC plus durvalumab and bevacizumab followed by SBRT for HCC.

To evaluate the safety of HAIC plus durvalumab and bevacizumab followed by SBRT for HCC.

Exploratory Objective(s):

Evaluate the consistency of imaging CR and pathological CR in resected patients, and explore biomarkers associated with prognosis .

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age > 18 years.
3. Have a HCC diagnosis confirmed by radiology, histology, or cytology.
4. HCC newly diagnosed or recurrent with a history of surgery or ablation, not amenable to curative surgery or transplantation.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to screening.
7. Tumours were classified as unresectable after a multidisciplinary team review because either:

   1. R0 resection was not feasible
   2. Sum of tumor diameters ≥5cm
   3. A maximum of three tumour lesions
   4. For patients with tumors located in bilateral hepatic lobes, the study requires that the number of tumors in the contralateral hepatic lobe of the larger tumor be less than 3, and the maximum tumor diameter should not exceed 3 cm.
8. Child-Pugh liver function score A.
9. Intrahepatic vascular invasion includes intrahepatic portal vein branch invasion, left or right portal vein invasion was allowed.
10. Patients with oligometastasis, defined as having a single metastatic organ with three or fewer metastases, each less than 3cm in size were permitted.
11. No prior radiotherapy or radioembolization to the liver or upper abdomen was allowed. Prior local therapies, such as surgery, radiofrequency ablation, percutaneous ethanol injection or cryoablation, are allowed if the index lesion(s) remain outside of the treatment field or have progressed since prior treatment. Local therapy must have been completed at least 4 weeks prior to the baseline scan.
12. Participants with HBV infection, characterized by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10 IU/ml or above the limit of detection per local lab standard), must be treated with antiviral therapy, as per institutional practice. Following antiviral therapy initiation, participants must show evidence of HBV stabilization or signs of viral response (eg, reduction HBV DNA levels) prior to study invention. Participants will remain on antiviral therapy for study duration and for 6 months after the last dose of study medication. Participants who test positive for anti HBV with undetectable HBV DNA (<10 IU/ml or under the limit of detection per local lab standard) do not require anti-viral therapy prior to enrollment. These subjects will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (≥10 IU/ml or above the limit of detection per local lab standard). HBV DNA detectable subjects must initiate and remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication.
13. Patients with active HCV infection as characterized by the presence of detectable HCV RNA upon enrollment must be managed per local institutional practice.
14. Life expectancy of >12 weeks.
15. Body weight >30 kg.
16. Adequate organ and marrow function, as defined below. Criteria "a," "b," "c," and "f" cannot be met with transfusions, infusions, or growth factor support administered within 14 days of starting the first dose.

    1. Hemoglobin ≥9 g/dL
    2. Absolute neutrophil count ≥1000/µL
    3. Platelet count ≥75000/µL
    4. Total bilirubin (TBL) ≤2.0× upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    5. AST and ALT ≤5×ULN
    6. Albumin ≥2.8 g/dL
    7. International normalized ratio (INR) ≤ 1.6. Note: INR prolongation due to anticoagulants for prophylaxis (e.g. atrial fibrillation) in patients without liver cirrhosis could be an exception
    8. Calculated creatinine clearance ≥40 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance
    9. 2+ proteinuria or lower urine dipstick reading. Participants having > 2+ proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥ 1 g/24 hours will be ineligible
17. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
18. Female participants:

    * Female participants must be 1 year post-menopausal, surgically sterile, or using one highly effective form of birth control (a highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly.) They should have been stable on their chosen method of birth control for a minimum of 3 months before entering the study.
    * Non-sterilized male partners of a woman of childbearing potential must use a male condom plus spermicide (condom alone in countries where spermicides are not approved) throughout this period.
    * Must show evidence of post-menopausal status or have a negative urinary or serum pregnancy test for female pre-menopausal patients.
19. Male Participants:

    * Male participants who intend to be sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable method of contraception from the time of screening throughout the total duration of the study and for drugs that are potentially genotoxic the drug washout period to prevent pregnancy in a partner.

Male participants must not donate or bank sperm during this same time period.

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma and HCC, or infiltrative-type HCC.
2. Intrahepatic or Extrahepatic vascular involvement: main hepatic vein invasion (VP3) or main portal vein (VP4).
3. Prior radiotherapy to the liver or upper abdomen.
4. Participation in another clinical study with an investigational product.
5. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
6. Receipt of the systematic anticancer therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, monoclonal antibodies) prior to the first dose of study drug.
7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the investigator.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the investigator.
8. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
9. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
11. History of allogenic organ transplantation.
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the investigator
    5. Patients with celiac disease controlled by diet alone
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
14. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
15. History of leptomeningeal carcinomatosis
16. History of active primary immunodeficiency
17. Confirmed HBV infection must not be co-infected with HCV (as indicated by the absence of anti-HCV antibodies) or hepatitis D virus (HDV: as indicated by the absence of anti-HDV antibodies).
18. Confirmed HCV infection must not be co-infected with HBV as defined by negative HBsAg. Patients with confirmed HCV infection who are negative for HBsAg, but positive for anti-HBV with detectable HBV DNA, are eligible but must be started on active antiviral therapy (for HBV) prior to enrollment to ensure adequate viral suppression (HBV DNA ≤2000 IU/mL).
19. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
20. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
21. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90days after the last dose of IP.
22. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
23. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
24. Prior treatment in a previous durvalumab clinical study regardless of treatment arm assignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | 3 MONTH

SECONDARY OUTCOMES:
Overall response rate (ORR) measured by RECIST v1.1, mRECIST. | 6 MONTH
Pathological complete response (pCR) for patients received resection. | 6 MONTH
Major pathologic response (MPR) for patients received resection. | 6 MONTH
AE | 6 MONTH

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China